CLINICAL TRIAL: NCT03409783
Title: A Multicenter Randomized Controlled Trial Evaluating the Effectiveness of the Enso Device for Treatment of Chronic Low Back Pain in Relation to Study Entry Criteria
Brief Title: Enso Pilot Study for Chronic Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to enroll into this study due to costs and other factors
Sponsor: Thimble Bioelectronics, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 17-02
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single blind, randomized, sham controlled study
Who Masked: Participant
Masking Description: Devices are assigned per the randomization schedule, with the sham device identical to the active device in every way except that no neuromodulation is delivered. The neuromodulation that the active device delivers can be done in a way that causes no sensation, so subjects are not unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active or ENSO Group (Active Comparator): Active ENSO device use for two weeks, at least one hour daily, including coaching via a smartphone app and coaching phone calls regarding device usage.
  Interventions: Device: ENSO Device
- Sham Group (Sham Comparator): Sham device use for two weeks, at least one hour daily, including coaching via a smartphone app and coaching phone calls regarding device usage.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: ENSO Device — An active ENSO device that delivers neuromodulation therapy.
  Arms: Active or ENSO Group
Device: Sham Device — Sham Device
  Arms: Sham Group

SUMMARY:
Enso is a portable device for the treatment of chronic and acute types of musculoskeletal pain. This study is being designed as a single blind, sham-controlled randomized clinical trial.

DETAILED DESCRIPTION:
Fifty subjects will be selected based on the inclusion criteria and then randomized to either the intervention group or the sham control group. Each subject will be randomly fitted with an Enso or a sham device and will be instructed to self-administer treatment daily for one hour or more per day for two weeks in both cohorts. Throughout the duration of the study, data will be recorded via a smartphone application regarding treatment usage and intensity, pain levels, the subject's impression of any changes in their functionality, and their opioid and non-opioid medication intake. Additional functional testing will be conducted at each study visit.

At the 2 week visit, the study blind will be broken, and subjects who were randomized to the sham group will be given the opportunity to cross over for an additional 2 week period using the active device.

ELIGIBILITY:
Inclusion Criteria:

1. Walk no further than 250 meters during a pre-study administration of the Six Minute Walk Test
2. Confirm that either they are able on their own to place the device (i.e., the gel pad) in its proper location, or they have a caretaker or family member who can assist them if needed
3. Mechanical (myofascial), axial back pain (focused around the spine)
4. 6/10 or greater level of pain
5. Functionally debilitated by their pain (e.g., difficulty walking)
6. Minimal radicular symptoms with no effect on functionality, medication, quality of life
7. Expressed desire to stop taking pain medications
8. Expressed desire to improve disability
9. 80% or greater of disability is due to pain in the low back (as opposed to other body areas)
10. Experiencing chronic pain for at least 6 months
11. Interested in being active, improving their functionality
12. Comfortable with using technology in daily life
13. Subject able to understand and grant informed consent
14. Documented adherence with clinic follow up visits per medical records
15. Has an email account
16. Above 18 years old

Exclusion Criteria:

1. Patients that do not own or have access to a smartphone
2. Subject who, in the Investigator's opinion, does not demonstrate a strong desire to reduce opioid or other pain medication usage (e.g., opioid dependence)
3. Has spinal instability, joint instability, or grade 2 or greater spondylolisthesis with instability
4. Primary symptoms due to spinal stenosis
5. Source of back pain related to an acute nerve impingement
6. Diagnosis of cancer/malignant tumors in the last 5 years
7. Source of back pain is an infection
8. Prior spinal fusion surgery
9. Has a cardiac pacemaker, implanted defibrillator or other implanted electronic device
10. Has radicular pain symptoms that account for more than 20% of their pain and/or functional impairment
11. Has undergone surgery to solve pain related to the study indication in the past 6 months
12. Patients with history of opioid, alcohol or drug abuse in the last 5 years, per investigator discretion
13. Any psychiatric condition that may interfere with the study assessments or prevent the subject from complying with the requirements of the protocol, in the judgement of the investigator.
14. Inability to complete subjective data as required; e.g. on mobile application and questionnaires
15. Pregnant women (as determined by self-report)
16. Have severe epilepsy
17. Have severe form of cardiovascular disease
18. Any other disease, condition, or habit(s) that in the opinion of the Principal Investigator would interfere with study compliance or adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Once a week for two weeks
  Compare the change in patient's 6 Minute Walk Test (6MWT) between the Enso intervention group and the sham group using the validated 6MWT procedure.

SECONDARY OUTCOMES:
Functional back pain assessment | Once a week for two weeks
  Functional back pain assessment using a 0 to 10 Numeric Pain Intensity Scale, assessed immediately after the 6MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Tay, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Spine and Nerve Diagnostic Center, Roseville, California
  - University of California, San Francisco, California

IPD SHARING:
Plan to Share IPD: No